CLINICAL TRIAL: NCT00384254
Title: Tobacco Quitlines as an Adjunct to Dental Office Tobacco Intervention
Brief Title: Tobacco Quitlines:Adjunct to Dental Office Tobacco Intervention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA 17972; R01DA017972 (NIH)
Record Dates: First submitted 2006-10-03; First posted 2006-10-06 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Tobacco Use Cessation
Keywords: Tobacco.; Cessation.; Dental patients.; Dentists.; Hygienists.; Dental assistants.; Health care providers.; Behavioral intervention.; Tobacco intervention.; Cigarettes.; Smokeless tobacco.; Smoking intervention.
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (No Intervention): Usual Care Control: Patients receive treatment as usual
- 2 (Experimental): "5 A" Intervention Condition: Patients in this condition receive all five "A" components (Ask, Advise, Assess, Assist, Arrange) recommended in the Clinical Practice Guideline: Treating Tobacco Use and Dependence.
  Interventions: Behavioral: 5 A
- 3 (Experimental): "3 A" Condition: Patients receive Ask, Advise, Arrange intervention consisting of the first two "A" components recommended by the Clinical Practice Guideline: Treating tobacco Use and Dependence, plus Fax-to-Quit referral to a tobacco quit line.
  Interventions: Behavioral: 3 A

INTERVENTIONS:
Behavioral: 5 A — Dental providers are trained to provide Ask, Advise, Assess, Assist and Arrange to all tobacco using patients. Written materials are provided, including information on local cessation resources, pharmacotherapy and tobacco quitlines.
  Arms: 2
Behavioral: 3 A — Providers are trained to provide Ask, Advise and Arrange intervention to all tobacco using patients. Written materials, prescription for NRT and a Fax-to-Quit referral are provided.
  Arms: 3

SUMMARY:
The purpose of the study is to compare two methods for providing brief dental office-based interventions designed to help patients quit either cigarette smoking or smokeless tobacco use, and to compare these two dental office-based interventions with usual care. This trial will evaluate the effectiveness of a unique combination of dental office intervention plus referral to the telephone help line, both of which have been demonstrated to be effective interventions for tobacco cessation. The integration of two lines of research-dental office interventions and telephone help line effectiveness-led us to propose this clinical trial as a more efficient and disseminable model of both training and practice.

DETAILED DESCRIPTION:
Although many dental practitioners now routinely incorporate the first two of the "5A's" (Ask and Advise) into their practice, and previous research indicates that brief office-based interventions are effective in producing modest tobacco quit rates for dental patients, dental practitioners continue to perceive a number of obstacles to routine provision of tobacco cessation services. Many dental practitioners still believe that counseling patients to quit an addictive behavior is beyond the scope of their training or comfort.

Recent studies have shown that proactive phone counseling from State-sponsored telephone tobacco help lines has a positive effect on tobacco cessation. The use of these help lines offers a unique supplement to the dental professional that could reduce the burden on practitioner and enhance the likelihood of their patients' quitting. Referral to a specialist is within the common heuristic followed by dental and medical practitioners. Therefore, we believe referral to a telephone help line may be an innovative way of enabling dentists and dental hygienists to encourage and support their patients to quit tobacco.

We will test two levels of intervention as compared to usual care in a randomized clinical trial in which 60 dental practices in Mississippi are randomized to one of three conditions. In one condition ("5A's"), the dental team will provide a brief office-based intervention that is modeled on the "5A's" advocated by the Clinical Practice Guideline. In the second condition ("3A's" + THL), the dental team will provide the first three "A's" (Ask, Advise, Assess), and then refer patients to the State-supported telephone help line for provision of the cessation counseling and follow-up support. In the third condition (Usual Care), volunteering practices will ask their patients only to complete our study surveys.

ELIGIBILITY:
Inclusion Criteria:

* Adult tobacco-using dental patients, aged 18 and older who come in for a regularly scheduled visit to a dentist or dental hygienist participating in our study.
* Dentists in private practice, employing at least one dental hygienist and one dental assistant.

Exclusion Criteria:

* Dental patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2177 (Actual)
Dates: Start 2004-01; Primary Completion 2007-11 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome is self-reported consecutive quit at 3 and 12 months following intervention. | 3 and 12 month
Secondary outcomes are reduction in use, number of quit attempts at 3 and 12 months, and increases in readiness to quit. | 3 and 12 months

SECONDARY OUTCOMES:
Conduct an economic analysis to determine the incremental cost per quit of the two interventions. | 12 month
Examine predictors of patient outcomes and the interaction of these variables with intervention condition. | 12 month
Examine patients' report of practitioner protocol delivery at six weeks as a function of intervention condition. | 6 week and 12 month
Examine the mediating effect of patient report of protocol delivery on patient outcomes across conditions. | 12 month
Assess practitioner report of implementation (at 3 months) and maintenance (at 12 months) of the protocol. | 3 and 12 month
Assess the effect of the intervention condition on changes in self-reported attitudes of dentists, dental hygienists, and dental assistants. | 3 and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Judith S. Gordon, Ph.D, Principal Investigator — Oregon Research Institute
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

REFERENCES:
- [Result] Gordon JS, Andrews JA, Crews KM, Payne TJ, Severson HH. The 5A's vs 3A's plus proactive quitline referral in private practice dental offices: preliminary results. Tob Control. 2007 Aug;16(4):285-8. doi: 10.1136/tc.2007.020271. PMID 17652247
- [Result] Gordon JS, Andrews JA, Crews KM, Payne TJ, Severson HH, Lichtenstein E. Do faxed quitline referrals add value to dental office-based tobacco-use cessation interventions? J Am Dent Assoc. 2010 Aug;141(8):1000-7. doi: 10.14219/jada.archive.2010.0314. PMID 20675426
- [Derived] Holliday R, Hong B, McColl E, Livingstone-Banks J, Preshaw PM. Interventions for tobacco cessation delivered by dental professionals. Cochrane Database Syst Rev. 2021 Feb 19;2(2):CD005084. doi: 10.1002/14651858.CD005084.pub4. PMID 33605440